CLINICAL TRIAL: NCT04054921
Title: An Open Label Extension Study of PTG-300 In Non-Transfusion Depenent (NTD) and Trasfusion-Dependent (TD) B-Thalassemia Subjects
Brief Title: Safety Study for Beta Thalassemia Subjects on PTG-300
Acronym: TRANSCEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTG-300-03
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-02

CONDITIONS: β-thalassemia; Ineffective Erythropoiesis
Keywords: Chronic anemia; β-thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventions (Experimental): PTG-300
  Interventions: Drug: PTG-300

INTERVENTIONS:
Drug: PTG-300 — PTG-300 is a hepcidin Mimetic

SUMMARY:
In this study will investigate long term safety and use of the PTG-300 in Beta Thalassemia patients.

DETAILED DESCRIPTION:
The PTG-300-03 study will study beta thalassemia patients on PTG-300 for two years. The dose and dose frequency for each subject enrolling in the PTG-300-03 study will be based on the last dose and frequency received by the subject in the previous study PTG-300-02 and the subject's response at that dose. Patients dose will be increased in a manner similar to that used on PTG-300-02 study. The maximum PTG-300 dose allowed is 80 mg/week.

ELIGIBILITY:
Inclusion Criteria:

* NTD and TD β-thalassemia subjects who completed Week 12 and Week 16 respectively in Study PTG-300-02.

Exclusion Criteria:

* Subjects who discontinued prematurely from study 300-02 (before Week 12 in NTD and Week 16 in TD).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with side effects and severity of side effects will be tabulated | Over two year Period after receiving PTG-300
  the long-term safety and tolerability of PTG-300 in Beta Thalassemia.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (2):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Boston Children's Hospital, Boston, Massachusetts
- Greece (3):
  - Laiko General Hospital of Athens, Athens
  - Athens General Hospital 'G Gennimatas', Athens
  - University General Hospital of Patras, Pátrai
- Chronic Care Center, Hazmiyeh, Lebanon
- Malaysia (2):
  - Hospital Ampang, Ampang
  - Hospital Umum Sarawak, Kuching
- Thailand (4):
  - Siriraj Hospital Mahidol University, Bangkok
  - Khon Kaen University, Khon Kaen
  - Chulalongkorn University, Pathum Wan
  - Naresuan University, Phitsanulok
- University Hospital Farhat Hached, Sousse, Tunisia
- Turkey (Türkiye) (2):
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No